CLINICAL TRIAL: NCT03981614
Title: Combination of MEK Inhibitor Binimetinib and CDK4/6 Inhibitor Palbociclib in KRAS and NRAS Mutant Metastatic Colorectal Cancers
Brief Title: Binimetinib and Palbociclib or TAS-102 in Treating Patients With KRAS and NRAS Mutant Metastatic or Unresectable Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-GI-1618; NCI-2019-03480 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-GI-1618 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Results first posted 2022-12-29 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Colorectal Carcinoma; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8; Unresectable Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — binimetinib; palbociclib; Trifluridine; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (binimetinib, palbociclib) (Experimental): Patients receive binimetinib PO BID on days 1-28 and palbociclib PO QD on days 1-21. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Binimetinib; Drug: Palbociclib
- Arm B (trifluridine and tipiracil hydrochloride) (Experimental): Patients receive trifluridine and tipiracil hydrochloride PO BID on days 1-5 and 8-12. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients with disease progression may optionally crossover to Arm A.
  Interventions: Drug: Trifluridine and Tipiracil Hydrochloride

INTERVENTIONS:
Drug: Binimetinib — Given PO
  Other Names: ARRY-162; ARRY-438162; MEK162; Mektovi
  Arms: Arm A (binimetinib, palbociclib)
Drug: Palbociclib — Given PO
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991
  Arms: Arm A (binimetinib, palbociclib)
Drug: Trifluridine and Tipiracil Hydrochloride — Given PO
  Other Names: Lonsurf; TAS 102; TAS-102; Tipiracil Hydrochloride Mixture with Trifluridine; Trifluridine/Tipiracil; Trifluridine/Tipiracil Hydrochloride Combination Agent TAS-102
  Arms: Arm B (trifluridine and tipiracil hydrochloride)

SUMMARY:
This phase II trial studies how well binimetinib and palbociclib work compared to TAS-102 in treating patients with KRAS and NRAS mutation positive colorectal cancer that has spread to other places in the body (metastatic) or cannot be removed by surgery (unresectable). Binimetinib and palbociclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as TAS-102, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving binimetinib and palbociclib may work better compared to TAS-102 alone in treating patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. The primary objective is to compare the progression-free survival (PFS) between those randomized to palbociclib/binimetinib and those randomized to trifluridine and tipiracil hydrochloride (TAS-102) in patients with refractory KRAS- or NRAS-mutant metastatic colorectal cancer (CRC).

SECONDARY OBJECTIVES:

I. To compare the overall response rate by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria between those randomized to palbociclib/binimetinib and those randomized to TAS-102 in patients with refractory KRAS- or NRAS-mutant metastatic CRC.

II. To compare the overall survival (OS) between those randomized to palbociclib/binimetinib and those randomized to TAS-102 in patients with refractory KRAS- or NRAS-mutant metastatic CRC.

III. To determine the safety and tolerability of the recommended phase II dose of palbociclib in combination with binimetinib in patients with refractory KRAS- or NRAS-mutant metastatic CRC.

CORRELATIVE RESEARCH OBJECTIVES:

I. To determine the tumor mutational profiles that characterize groups of patients that predict for response or resistance to combination of palbociclib/binimetinib.

II. To determine the correlation between circulating tumor deoxyribonucleic acid (DNA) and tumor response or resistance to therapy with palbociclib/binimetinib or TAS-102.

III. To determine the association between Consensus Molecular Subtype based on gene expression profiling and response or resistance to combination of palbociclib/binimetinib.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive binimetinib orally (PO) twice daily (BID) on days 1-28 and palbociclib PO once daily (QD) on days 1-21. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive trifluridine and tipiracil hydrochloride PO BID on days 1-5 and 8-12. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients with disease progression may optionally crossover to Arm A.

After completion of study treatment, patients are followed up within 30-37 days and then every 12 weeks for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of colorectal cancer that is metastatic and/or unresectable
* Documented mutation in KRAS or NRAS (codon 12, 13, 59, 61, 117, or 146) in tumor tissue from primary or metastatic site, tested by a Clinical Laboratory Improvement Act (CLIA)-certified laboratory
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Previously treated with fluoropyrimidine, oxaliplatin, and irinotecan based chemotherapy, and an anti-VEGF biological therapy
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (obtained =< 14 days prior to registration/randomization unless otherwise noted)
* Platelet count >= 75 x 10^9/L without transfusions (obtained =< 14 days prior to registration/randomization unless otherwise noted)
* Hemoglobin (Hgb) >= 9 g/dL (obtained =< 14 days prior to registration/randomization unless otherwise noted)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration/randomization unless otherwise noted)
* Aspartate transaminase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN; =< 5.0 x ULN if known liver metastases (obtained =< 14 days prior to registration/randomization unless otherwise noted)
* Serum creatinine =< 1.5 mg/dL OR calculated creatinine clearance >= 50 mL/min using the Cockcroft-Gault formula (obtained =< 14 days prior to registration/randomization unless otherwise noted)
* Negative serum beta-human chorionic gonadotropin (B-HCG) pregnancy test done =< 7 days prior to registration/randomization for women of childbearing potential only
* Able to swallow capsules with no surgical or anatomic conditions that would preclude the patient from swallowing and absorbing oral medications
* Able and willing to provide informed written consent and able to comply with protocol requirement
* Able and willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

  * NOTE: During the active monitoring phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* Willing to provide blood and tissue samples for mandatory correlative research purposes
* Patient is deemed by the investigator to have the initiative and means to be compliant with the protocol (treatment and follow-up)
* CROSSOVER INCLUSION CRITERIA: Histological confirmation of colorectal cancer that is metastatic and/or unresectable
* CROSSOVER INCLUSION CRITERIA: Documented mutation in KRAS or NRAS (codon 12, 13, 59, 61, 117, or 146) in tumor tissue from primary or metastatic site, tested by a CLIA-certified laboratory
* CROSSOVER INCLUSION CRITERIA: Measurable disease
* CROSSOVER INCLUSION CRITERIA: ECOG performance status (PS) of 0 or 1
* CROSSOVER INCLUSION CRITERIA: Previously treated with fluoropyrimidine, oxaliplatin, and irinotecan based chemotherapy, and an anti-VEGF biological therapy
* CROSSOVER INCLUSION CRITERIA: ANC >= 1.5 x 10^9/L (obtained =< 28 days of re-registration unless otherwise noted)
* CROSSOVER INCLUSION CRITERIA: Platelet count >= 75 x 10^9/L without transfusion (obtained =< 28 days of re-registration unless otherwise noted)
* CROSSOVER INCLUSION CRITERIA: Hgb >= 9 g/dL (obtained =< 28 days of re-registration unless otherwise noted)
* CROSSOVER INCLUSION CRITERIA: Total bilirubin =< 1.5 x ULN (obtained =< 28 days of re-registration unless otherwise noted)
* CROSSOVER INCLUSION CRITERIA: AST and ALT =< 2.5 x ULN; =< 5.0 x ULN if known liver metastases (obtained =< 28 days of re-registration unless otherwise noted)
* CROSSOVER INCLUSION CRITERIA: Serum creatinine =< 1.5 mg/dL OR calculated creatinine clearance >= 50 mL/min using the Cockcroft-Gault formula (obtained =< 28 days of re-registration unless otherwise noted)
* CROSSOVER INCLUSION CRITERIA: Negative serum beta-HCG pregnancy test done =< 7 days prior to re-registration for women of childbearing potential only
* CROSSOVER INCLUSION CRITERIA: Able to swallow capsules with no surgical or anatomic conditions that would preclude the patient from swallowing and absorbing oral medications
* CROSSOVER INCLUSION CRITERIA: Able and willing to provide informed written consent and able to comply with protocol requirements
* CROSSOVER INCLUSION CRITERIA: Able and willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

  * NOTE: During the Active Monitoring phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* CROSSOVER INCLUSION CRITERIA: Willing to provide blood samples for mandatory correlative research purposes
* CROSSOVER INCLUSION CRITERIA: Patient is deemed by the investigator to have the initiative and means to be compliant with the protocol (treatment and follow-up)

Exclusion Criteria:

* Prior treatment with drug targeting BRAF, MEK, ERK, or CDK family

  * NOTE: For the purpose of this protocol, prior treatment with regorafenib is allowed
* Prior treatment with trifluridine/tipiracil (TAS-102)
* Pregnant or nursing (lactating women), where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
* Women of child-bearing potential

  * NOTE: defined as all women physiologically capable of becoming pregnant, unless they agree to use highly effective methods of contraception throughout the study and for 8 weeks after study drug discontinuation
  * NOTE: Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation >= 42 days prior to registration/randomization. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of child bearing potential
* Sexually active males

  * NOTE: unless they agree to use highly effective methods of contraception throughout the study and for 12 weeks after study drug discontinuation and should not father a child in this period
* Any symptomatic brain metastasis

  * NOTE: Patients previously treated or untreated for this condition who are asymptomatic in the absence of corticosteroid and anti-epileptic therapy are allowed. Brain metastases must be stable for >= 4 weeks prior to registration/randomization, with imaging (e.g., magnetic resonance imaging [MRI] or computed tomography [CT]) demonstrating no current evidence of progressive brain metastases at registration/randomization
* Prior treatment =< 21 days prior to registration/randomization with any other chemotherapy, small molecule inhibitor (e.g. regorafenib), monoclonal antibody, immunotherapy, or radiotherapy

  * NOTE: All toxicities from prior therapy must be =< grade 1 (or =< grade 2 for peripheral neuropathy or alopecia)
* Impaired cardiovascular function or clinically significant cardiac diseases, including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) < 6 months prior to registration/randomization
  * Symptomatic chronic heart failure (i.e. grade 2 or higher), history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality < 6 months prior to registration/randomization except atrial fibrillation and paroxysmal supraventricular tachycardia
  * Left ventricular ejection fraction (LVEF) < 50% as determined by a multigated acquisition (MUGA) scan or echocardiogram =< 28 days prior to registration/randomization
* Uncontrolled hypertension, defined as persistent elevation of systolic blood pressure >= 150 mmHg or diastolic blood pressure >= 100mmHg despite current therapy
* History of thromboembolic or cerebrovascular events =< 12 weeks prior registration/randomization. Examples include transient ischemic attacks, cerebrovascular accidents, hemodynamically significant (i.e. massive or submassive) deep vein thrombosis or pulmonary emboli

  * Note: Patients with either deep vein thrombosis or pulmonary emboli that does not result in hemodynamic instability are allowed to enroll as long as they are on a stable dose of anticoagulants for at least 4 weeks
  * Note: Patients with thromboembolic events related to indwelling catheters or other procedures may be enrolled
* Known history of acute or chronic pancreatitis =< 6 months prior to registration/randomization
* Known positive serology for HIV (human immunodeficiency virus), active hepatitis B, and/or active hepatitis C infection
* Patients who have neuromuscular disorders that are associated with elevated creatine phosphokinase (CPK) (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* History of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) =< 12 months prior to registration/randomization
* Impaired gastrointestinal (GI) function or disease that may significantly alter the absorption of binimetinib or palbociclib (e.g., ulcerative disease, uncontrolled vomiting, malabsorption syndrome, small bowel resection with decreased intestinal absorption) in the opinion of the investigator
* History or current evidence of retinal vein occlusion (RVO) or current risk factors to RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes)
* Leptomeningeal disease
* Known hypersensitivity to the components of study drugs or its analogs
* Known medical, psychiatric, substance abuse, or cognitive disorder that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements in the opinion of the investigator
* Patients who have undergone major surgery =< 21 days prior to registration/randomization or who have not recovered from side effects of such procedures
* Any other co-morbid, systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Previous or concurrent malignancy =< 3 years prior to registration/randomization with the following exceptions:

  * Adequately treated basal cell or squamous cell carcinoma of the skin
  * Superficial bladder cancer
  * Prostate intraepithelial neoplasm
  * In situ carcinoma of the cervix
  * Other solid tumors treated curatively without evidence of recurrence for >= 3 years prior to registration/randomization

    * NOTE: If there is a history or prior malignancy, must not be receiving other specific anti-cancer treatment such as anti-estrogen, anti-androgen, or other tyrosine kinase inhibitor therapy
* CROSSOVER EXCLUSION CRITERIA: Prior treatment with drug targeting BRAF, MEK, ERK, or CDK family

  * NOTE: For the purpose of this protocol, prior treatment with regorafenib is allowed
* CROSSOVER EXCLUSION CRITERIA: Pregnant or nursing (lactating women), where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
* CROSSOVER EXCLUSION CRITERIA: Women of child-bearing potential

  * NOTE: Defined as all women physiologically capable of becoming pregnant, unless they agree to use highly effective methods of contraception throughout the study and for 8 weeks after study drug discontinuation
  * NOTE: Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation >= 42 days of re-registration. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of child bearing potential
* CROSSOVER EXCLUSION CRITERIA: Sexually active males

  * NOTE: unless they agree to use highly effective methods of contraception throughout the study and for 12 weeks after study drug discontinuation and should not father a child in this period
* CROSSOVER EXCLUSION CRITERIA: Any symptomatic brain metastasis

  * NOTE: Patients previously treated or untreated for this condition who are asymptomatic in the absence of corticosteroid and anti-epileptic therapy are allowed. Brain metastases must be stable for >= 4 weeks, with imaging (e.g., MRI or CT) demonstrating no current evidence of progressive brain metastases at re-registration
* CROSSOVER EXCLUSION CRITERIA: Impaired cardiovascular function or clinically significant cardiac diseases, including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) < 6 months prior to re-registration
  * Symptomatic chronic heart failure (i.e., grade 2 or higher), history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality < 6 months prior to re-registration except atrial fibrillation and paroxysmal supraventricular tachycardia
  * Left ventricular ejection fraction (LVEF) < 50% as determined by a MUGA scan or echocardiogram
* CROSSOVER EXCLUSION CRITERIA: Uncontrolled hypertension, defined as persistent elevation of systolic blood pressure >= 150 mmHg or diastolic blood pressure >= 100 mmHg despite current therapy
* CROSSOVER EXCLUSION CRITERIA: History of thromboembolic or cerebrovascular events =< 12 weeks prior re-registration. Examples include transient ischemic attacks, cerebrovascular accidents, hemodynamically significant (i.e. massive or sub-massive) deep vein thrombosis or pulmonary emboli

  * Note: Patients with either deep vein thrombosis or pulmonary emboli that does not result in hemodynamic instability are allowed to enroll as long as they are on a stable dose of anticoagulants for at least 4 weeks
  * Note: Patients with thromboembolic events relat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kopetz, Principal Investigator — Academic and Community Cancer Research United
Locations (7):
- United States (7):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Binimetinib, Palbociclib): Patients receive binimetinib PO BID on days 1-28 and palbociclib PO QD on days 1-21. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  >
  >
  >
  >
  >
  > Binimetinib: Given PO
  >
  >
  >
  >
  >
  > Palbociclib: Given PO
- Arm B (Trifluridine and Tipiracil Hydrochloride): Patients receive trifluridine and tipiracil hydrochloride PO BID on days 1-5 and 8-12. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients with disease progression may optionally crossover to Arm A.
  >
  >
  >
  >
  >
  > Trifluridine and Tipiracil Hydrochloride: Given PO
- Safety Run-In Cohort: In the safety run-in, an initial cohort will receive palbociclib orally once daily on days 1-21 out of a 28 day cycle and binimetinib orally twice per day continuously at 30 mg BID daily. The starting dose of palbociclib will be 100 mg orally once daily on days 1-21 out of a 28 day cycle. If the starting dose is not well tolerated, with 2 or more subjects experiencing excessive toxicity as defined in Section 7.15, then the dose will be reduced to 75 mg orally once daily on days 1-21 out of a 28 day cycle dose, and further de-escalation will be studied if needed to determine a safe and tolerable dose in this population of colorectal cancer patients.
Period: Overall Study
Arm/Group | Arm A (Binimetinib, Palbociclib) | Arm B (Trifluridine and Tipiracil Hydrochloride) | Safety Run-In Cohort
Started | 47 | 46 | 9
Crossed Over to Arm A | 0 | 21 | 0
Completed | 42 | 41 | 8
Not Completed | 5 | 5 | 1
Not completed — Patient withdrawn prior to treatment | 5 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A (Binimetinib, Palbociclib): Patients receive binimetinib PO BID on days 1-28 and palbociclib PO QD on days 1-21. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.>> >> Binimetinib: Given PO>>
  >> Palbociclib: Given PO
- Arm B (Trifluridine and Tipiracil Hydrochloride): Patients receive trifluridine and tipiracil hydrochloride PO BID on days 1-5 and 8-12. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients with disease progression may optionally crossover to Arm A.>>
  >> Trifluridine and Tipiracil Hydrochloride: Given PO
- Total: Total of all reporting groups
Arm/Group | Arm A (Binimetinib, Palbociclib) | Arm B (Trifluridine and Tipiracil Hydrochloride) | Safety Run-In Cohort | Total
Number analyzed (Participants) | 42 | 41 | 8 | 91
Age, Continuous [Median (Full Range); unit: years] | 52 [32 to 73] | 52 [33 to 74] | 51.5 [43 to 68] | 52 [32 to 74]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 19 | 22 | 3 | 44
  Gender: Female | 23 | 19 | 4 | 46
  Gender: Unknown | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 0 | 5
  White | 41 | 32 | 6 | 79
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 42 | 41 | 8 | 91
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG performance status evaluates a patient's ability to perform every-day tasks; a higher score is associated with more impairment.>> 0 - Fully active, able to carry on all pre-disease performance without restriction>>
  1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    0 | 19 | 19 | 5 | 43
    1 | 23 | 22 | 3 | 48

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Disease progression will be determined based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and will be documented at each enrolling site with no central review planned. PFS will be compared between treatment arms using the stratified log rank test at one-sided level 0.05. Kaplan-Meier methodology will be used to estimate the median PFS for each treatment arm, and Kaplan-Meier curves will be produced.
Time Frame: Time from randomization date to either disease progression or death from any cause, whichever occurs first, assessed for up to 16 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm A (Binimetinib, Palbociclib): Patients receive binimetinib PO BID on days 1-28 and palbociclib PO QD on days 1-21. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.> >>
  >
  >> Binimetinib: Given PO>
  >>
  >
  >> Palbociclib: Given PO
- Arm B (Trifluridine and Tipiracil Hydrochloride): Patients receive trifluridine and tipiracil hydrochloride PO BID on days 1-5 and 8-12. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients with disease progression may optionally crossover to Arm A.>
  >>
  >
  >> Trifluridine and Tipiracil Hydrochloride: Given PO
Arm/Group | Arm A (Binimetinib, Palbociclib) | Arm B (Trifluridine and Tipiracil Hydrochloride)
Number analyzed (Participants) | 42 | 41
months | 2.3 [2.0 to 3.0] | 2.2 [2.1 to 2.3]

2. Secondary Outcome: Overall Response Rate
Description: Assessment of response data will be performed on the basis of definitions of responses according to RECIST version (v)1.1. Objective response is defined as a complete or partial response by RECIST v1.1. This will be reported as the number of patients experiencing an objective response.
Time Frame: Up to 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Binimetinib, Palbociclib) | Arm B (Trifluridine and Tipiracil Hydrochloride)
Number analyzed (Participants) | 42 | 41
Participants | 0 | 1

3. Secondary Outcome: Overall Survival (OS)
Description: Will use Kaplan-Meier methods to evaluate time to event endpoints, and will report median OS and its 95% confidence interval.
Time Frame: Time from first dose of study treatment to death from any cause, assessed for up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Binimetinib, Palbociclib) | Arm B (Trifluridine and Tipiracil Hydrochloride)
Number analyzed (Participants) | 42 | 41
months | 7.7 [5.1 to 13.1] | 6.8 [5.5 to 8.4]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: The number of patients experiencing a grade 3+ adverse event, regardless of attribution, will be reported.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Binimetinib, Palbociclib) | Arm B (Trifluridine and Tipiracil Hydrochloride) | Safety Run-In Cohort
Number analyzed (Participants) | 42 | 41 | 8
Participants | 25 | 28 | 6

ADVERSE EVENTS:
Time Frame: 24 months
Groups:
- Crossover: After completion of treatment with Trifluridine and Tipiracil Hydrochloride: Given PO, patients were given the option of being treated with Palbociclib: Given PO, crossing over from arm B to arm A.
Arm/Group | Arm A (Binimetinib, Palbociclib) | Arm B (Trifluridine and Tipiracil Hydrochloride) | Crossover | Safety Run-In Cohort
All-Cause Mortality (participants affected / at risk) | 29/42 | 18/41 | 15/21 | 1/8
Serious Adverse Events (participants affected / at risk) | 9/42 | 12/41 | 5/21 | 4/8
Other Adverse Events (participants affected / at risk) | 38/42 | 39/41 | 21/21 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Binimetinib, Palbociclib) (N=42) | Arm B (Trifluridine and Tipiracil Hydrochloride) (N=41) | Crossover (N=21) | Safety Run-In Cohort (N=8)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CPK increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin T increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Binimetinib, Palbociclib) (N=42) | Arm B (Trifluridine and Tipiracil Hydrochloride) (N=41) | Crossover (N=21) | Safety Run-In Cohort (N=8)
Anemia (Blood and lymphatic system disorders) | 17 (28) | 26 (46) | 17 (30) | 6 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 3 (3) | 0 (0) | 3 (4) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (4)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 1 (2) | 0 (0) | 2 (3) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (5) | 2 (5) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (8) | 10 (16) | 7 (10) | 2 (3)
Anal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (7) | 6 (7) | 4 (6) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 13 (33) | 10 (14) | 8 (11) | 5 (10)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (3) | 2 (7) | 1 (2) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (6) | 5 (8) | 3 (5) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 2 (7) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 7 (14) | 0 (0) | 4 (6) | 2 (7)
Nausea (Gastrointestinal disorders) | 13 (22) | 15 (29) | 9 (10) | 4 (10)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (2) | 2 (3) | 1 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (15) | 12 (24) | 6 (8) | 3 (6)
Chills (General disorders) | 2 (3) | 1 (1) | 1 (2) | 2 (2)
Edema face (General disorders) | 1 (3) | 0 (0) | 1 (2) | 1 (3)
Edema limbs (General disorders) | 6 (15) | 5 (12) | 4 (9) | 3 (7)
Fatigue (General disorders) | 18 (45) | 13 (32) | 13 (17) | 5 (10)
Fever (General disorders) | 4 (5) | 0 (0) | 2 (2) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neck edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (2) | 2 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (9) | 6 (6) | 4 (7) | 3 (6)
Alkaline phosphatase increased (Investigations) | 11 (14) | 13 (26) | 9 (16) | 5 (8)
Aspartate aminotransferase increased (Investigations) | 10 (15) | 9 (13) | 7 (12) | 4 (6)
Blood bilirubin increased (Investigations) | 4 (5) | 9 (13) | 2 (2) | 1 (1)
CPK increased (Investigations) | 15 (38) | 0 (0) | 7 (11) | 6 (12)
Cardiac troponin I increased (Investigations) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Cardiac troponin T increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (4)
Cholesterol high (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 3 (3) | 1 (1) | 3 (6) | 1 (2)
Investigations - Other, specify (Investigations) | 3 (5) | 2 (4) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 7 (9) | 12 (17) | 5 (8) | 3 (5)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 15 (35) | 22 (37) | 8 (14) | 2 (4)
Platelet count decreased (Investigations) | 18 (37) | 10 (26) | 6 (8) | 6 (12)
Weight gain (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (2) | 0 (0) | 3 (3) | 0 (0)
White blood cell decreased (Investigations) | 16 (29) | 16 (40) | 5 (11) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 7 (9) | 7 (9) | 5 (10) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (6) | 1 (7) | 2 (3) | 1 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (12) | 7 (13) | 5 (8) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (6) | 2 (2) | 3 (3) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 3 (6) | 2 (3) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (6) | 3 (6) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 4 (7) | 1 (2) | 2 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 3 (5) | 4 (9) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (9) | 2 (4) | 1 (2) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 1 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3) | 2 (2) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (2) | 1 (2) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Concentration impairment (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 1 (1) | 3 (6) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5) | 4 (6) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (7) | 3 (7) | 2 (3) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (2) | 4 (13) | 2 (4) | 3 (6)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (2) | 1 (4) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 7 (10) | 3 (4) | 1 (1) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (2) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 5 (5) | 3 (4) | 2 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (11) | 6 (9) | 3 (4) | 3 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 1 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (3)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (5) | 1 (1) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 23 (48) | 2 (4) | 10 (19) | 7 (15)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (14) | 1 (1) | 2 (2) | 4 (6)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 6 (10) | 6 (11) | 4 (5) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT03981614/Prot_SAP_000.pdf